CLINICAL TRIAL: NCT04144660
Title: "Treatment Use of ECMO In Pregnancy or Peripartum Patient."
Status: Completed | Type: Observational
Sponsor: Sarah Thordsen (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Sarah Thordsen, Assistant Professor Cardiovascular Medicine, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Other Study IDs: PRO00036221
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Cardiogenic Shock; Peripartum Cardiomyopathy; Complication, Pregnancy
MeSH Terms: conditions — Shock, Cardiogenic; Peripartum Cardiomyopathy; Pregnancy Complications | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiogenic Shock Treated with ECMO: This cohort of participants required clinical intervention with ECMO for treatment of their index cardiogenic shock episode while pregnant or post delivery of their infant.
  Interventions: Device: Extracorporeal Membrane Oxygenation

INTERVENTIONS:
Device: Extracorporeal Membrane Oxygenation — Use of ECMO for circulatory / hemodynamic support of peripartum of pregnant patients who developed cardiogenic shock.

SUMMARY:
The goal of this study is to describe the use of ECMO (Extracorporeal Membrane Oxygenation) in the pregnant or peripartum patient.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18 years or greater at the time of ECMO treatment.
3. Pregnant or within 6 months post-partum at the time of ECMO cannulation

Exclusion Criteria:

1. No history of pregnancy.
2. No treatment with ECMO.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women treated with ECMO while pregnant or immediately postpartum (within six months).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome of Mother | Time of diagnosis -Six Month Survival Rate
  Describe clinical course of pregnant or recently postpartum patients with cardiogenic shock treated with ECMO, including the rate of neonate survival

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Thordsen, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided